CLINICAL TRIAL: NCT00406874
Title: Effect of Omega 3 Fats on Sperm Quality and Sexual Function in Infertile Men Age 35-55
Brief Title: Effect of Omega 3 Fats on Sperm Quality and Sexual Function
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: reports indicating that increased folic acid intake may increase colin cancer
Sponsor: Reproductive Partners Medical Group (Other)
Responsible Party: Principal Investigator, David R. Meldrum, M.D., Scientific Director, Reproductive Partners Medical Group
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPMG-1
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Infertility
Keywords: infertility; semen quality; sexual function; blood pressure; omega 3 fats; folic acid
MeSH Terms: conditions — Infertility | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: omega 3 fats — 1,000 mg daily
Drug: folic acid — 800 micrograms daily

SUMMARY:
This study compares the effects of omega 3 fats plus folic acid with placebo plus folic acid on sperm quality and sexual function in infertile men. It will also evaluate the effects on sexual fuction of a sub-therapeutic dose of a PDE 5 inhibitor versus placebo in subjects continuing on both omega 3 fats and folic acid.

DETAILED DESCRIPTION:
Infertile men commonly have difficulty timing sexual relations around the time of ovulation. There is a high incidence of abnormal sperm morphology in infertile men. Omega 3 fats are known to increase the production of nitric oxide, which is the mediator of the male response, and folic acid is an important cofactor in the production of nitric oxide. Omega 3 fats are also important in the structure and function of cell membranes. There is a high incidence of deficient intake of omega 3 fats and folic acid in the U.S. population. Both folic acid and omega 3 fats are available as nutritional supplements and the doses used in this study are doses commonly recommended as nutritional supplements.

Comparison: Omega 3 fats plus folic acid will be compared with placebo plus folic acid in men age 35 to 55 attempting pregnancy with normal or mildly impaired semen quality. They will fill out dietary questionaires, questionaires regarding sexual function, and will have measurements of serum nitrates, blood pressure, and semen quality before and during use of these nutritional supplements. In men continuing on both omega 3 fats and folic acid, we will compare the effects of a sub-therapeutic dose of a PDE 5 inhibitor versus placebo on their sexual function.

ELIGIBILITY:
Inclusion Criteria:

* infertile men
* age 35 to 55
* expressing difficulty timing relations to their partner's ovulation

Exclusion Criteria:

* hypertension, heart disease or other systemic diseases
* fatty fish intake more than twice per week
* marked semen abnormalities (less than 10 million sperm per ml, less than 20 % A plus B motility, more than 1 million WBC per HPF)
* use of anticoagulants
* must be willing to not take PDE 5 inhibitors during the study
* use of other supplements is prohibited during the study

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Questionaires regarding sexual function | every 30 days
Semen analysis | every 30 days

SECONDARY OUTCOMES:
blood pressure | every 30 days
serum nitrate levels | every 30 days

CONTACTS AND LOCATIONS:
Overall Officials: David R Meldrum, M.D., Principal Investigator — Reproductive Partners Medical Group
Locations (1):
- Reproductive Partners medical Group, Redondo Beach, California, United States